CLINICAL TRIAL: NCT00467506
Title: Phase II Two-step Radioimmunotherapy Clinical Study in Medullary Thyroid Carcinoma
Acronym: RIT in MTC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: BRD 03/2-U
Record Dates: First submitted 2007-04-27; First posted 2007-04-30 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2011-11

CONDITIONS: Thyroid Neoplasms
Keywords: Recurrence of medullary thyroid carcinoma: abnormal calcitonin level and biomarkers doubling time lower than 5 years after initial surgery
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Antibodies, Bispecific

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: bispecific antibody and di-DTPA-131I

SUMMARY:
Phase II clinical trial assessing efficacy and toxicity of pretargeted radioimmunotherapy using anti-CEAxanti-DTPA bispecific antibody and di-DTPA-131I peptide in patients with reccurrence of medullary thyroid carcinoma (abnormal calcitonin level and biomarkers doubling time lower than 5 years)

ELIGIBILITY:
Inclusion Criteria:

* 18 -75 years
* Karnofsky ≥ 70%
* Histological diagnosis of medullary thyroid carcinoma
* Calcitonin serum level Ê 100 pg/ml and Calcitonin or CEA doubling time £ 5 years
* Normal liver and renal functions
* Granulocytes ≥ 1500/mm3 and platelets ≥ 150 000/mm3
* No immunization
* Consent form signed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francoise Bodere, MD, Principal Investigator — Nantes University Hospital
Locations (11):
- France (11):
  - Centre François Baclesse, Caen
  - CHU de Grenoble, Grenoble
  - hôpital du Cluzeau, Limoges
  - CHU, Lyon
  - Hôpital de la timone, Marseille
  - CHU, Nantes
  - CHU, Rouen
  - Centre René Huguenin, Saint-Cloud
  - Centre René Gauducheau, Saint-Herblain
  - Centre Paul Strauss, Strasbourg
  - Centre Claudius Régaud, Toulouse